CLINICAL TRIAL: NCT04165499
Title: Preliminary Study of Nutritional Intervention, Randomized, Double Blind, and Controlled Parallel Groups to Evaluate the Effect of Consuming a Combination of of Plant Extracts (BSL_EP026) on Serum Uric Acid in Hypeuricemic Subjects.
Brief Title: Effect of the Consumption of a Combination of Plant Extracts (BSL_EP026) on Serum Uric Acid.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Collaborators: Clínica Dr. Miguel Quesada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C026
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2019-07

CONDITIONS: Hyperuricemia
Keywords: Hyperuricemia; Plant extracts
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of Plant Extracts (BSL_EP026) (Experimental): Volunteers will take 1 capsule twice daily with the combination of the plant extracts (BSL_EP026).
  Interventions: Combination Product: Combination of Plant Extracts (BSL_EP026)
- Control (Placebo Comparator): Volunteers will take 1 capsule twice daily with maltodextrin.
  Interventions: Combination Product: Control

INTERVENTIONS:
Combination Product: Combination of Plant Extracts (BSL_EP026) — Each participant will consume 2 capsules daily, in the morning and in the evening.
  Arms: Combination of Plant Extracts (BSL_EP026)
Combination Product: Control — Each participant will consume 2 capsules daily, in the morning and in the evening.
  Other Names: Placebo group
  Arms: Control

SUMMARY:
The objective of this study is to evaluate the effect of the combination of a combination of plant extracts (BSL_EP026) on blood and urine uricemia levels in individuals with levels at the limit of the values considered normal or moderately high.

DETAILED DESCRIPTION:
Hyperuricemia is an abnormally high level of uric acid in the blood, resulted because of an increased production of uric acid, decreased excretion of uric acid, or both. This can cause gout and nephrolithiasis, and it has also been related to metabolic syndrome, diabetes mellitus, cardiovascular disease and chronic kidney disease.

Some plant extracts have diuretic activity that could contribute to improve uric acid excretion. This effect would lead to a decrease in uric acid plasma levels and, secondarily, to an action on its metabolic pathway of endogenous biogeneration.

On the other hand, uric acid has a double reabsorption-elimination step in the renal tubules and the flavonoids of both extracts impede the processes of renal resorption promoting urinary elimination, in addition to increase the pH of the urine (higher than pH 5.8), which favors the non-precipitation or formation of urate stones.

Finally, the routine (present in the used extracts) inhibit the uric acid formation pathway from purines, which would act synergistically.

In this project, the effect of the intake of a combination plant extracts on uricemia levels will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Blood uric acid levels greater than 7 mg/dL in men and 6 mg dL in women.
* Accept freely to participate in the study and sign the informed consent document.

Exclusion Criteria:

* Having treatment that can affect uric acid levels.
* Use of diuretics.
* Follow a low purine diet.
* Take a food supplement or drug that interferes with uric acid metabolism and renal system function.
* Have an allergy to birch and/or orthosiphon or another component of the test products.
* Low compliance expectation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Uric acid | 2 weeks
  Uric acid in plasma

SECONDARY OUTCOMES:
Uric acid in urine | 2 weeks
  Uric acid in morning spot urine
pH of urine | 2 weeks
  pH in morning spot urine
Blood pressure | 2 weeks
  Systolic and diastolic pressure during the study
Fractional clearance of urate (FCU) | 2 weeks
  Renal clearance of urate/Renal clearance of creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Quesada, MD, PhD, Principal Investigator — Clínica Dr. Quesada
Locations (1):
- Biosearch Life, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No